CLINICAL TRIAL: NCT03202160
Title: Cases of Goiter in Children Attending Assiut University Children Hospital
Brief Title: Causes of Goiter in Children Attending Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MAAta, principal investigator, Assiut University
Other Study IDs: CGCA
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Goiter
Keywords: Goiter
MeSH Terms: conditions — Goiter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thyroid disorders are one of the most common endocrine problems in children and adolescents. Diagnostic considerations can be approached from the perspective of the goiter.A goiter, or thyromegaly, is an enlargement of the thyroid gland.Persons with enlarged thyroids can have normal function of the gland (euthyroidism), thyroid deficiency (hypothyroidism), or overproduction of the hormones (hyperthyroidism).

DETAILED DESCRIPTION:
Congenital goiter most commonly occurs in neonates born to mothers with known thyroid disease especially Graves' disease. Other causes of congenital goitrous hypothyroidism are thyroid dyshormonogenesis, endemic iodine deficiency and maternal goitrogen ingestion or iodine excess (expectorants, povidone iodine).

The most common causes of euthyroid goiter in childhood are chronic lymphocytic thyroiditis and a colloid goiter (simple goiter). Thyroid enlargement that is not caused by inflammatory, infectious or neoplastic causes is termed a colloid goiter, also.

Chronic lymphocytic thyroiditis , also known as Hashimoto thyroiditis, is an autoimmune, inflammatory process that causes up to 55% to 65% of all euthyroid goiters, and almost all cases of thyroiditis in childhood and adolescence. A large North American prevalence study showed that as many as 1.2% of children aged 11 to18 years have chronic lymphocytic thyroiditis, as defined by an enlarged thyroid gland and detectable serum thyroid antibodies.

Thyroid nodules are relatively common in adolescents; these nodules are usually asymptomatic and often discovered incidentally, but they raise the fear of cancer. A multi-nodular goiter is almost invariably caused by Hashimoto's thyroiditis and it carries a good prognosis. The asymptomatic, solitary thyroid nodule is a thyroid adenoma, thyroid carcinoma or a thyroid cyst. Thyroid carcinoma occurs in approximately one per one million persons/year in the first-two decades of life.

No reported data are found as regard of causes of goiter in children in our locality.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes of ages since birth up to 18 years old who are presented by goiter.

Exclusion Criteria:

* Any patient with neck swelling other than goiter.
* Refusal of participation.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All cases of goiter attending Assiut University hospitals of ages since birth up to 18 years old in the period of study
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Serum T3 and T4 | 1 day
  Serum T3 and T4 for diagnosis of cause of goiter
Neck ultrasonography | 1 day
  Neck ultrasonography for confirmation of diagnosis of goiter and for diagnosis of cause of goiter

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa A Mohammed, MD, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muirhead S. Diagnostic approach to goitre in children. Paediatr Child Health. 2001 Apr;6(4):195-9. doi: 10.1093/pch/6.4.195. PMID 20084235